CLINICAL TRIAL: NCT05654233
Title: The Study of Reducing Adverse Effects After Radiofrequency Ablation Combined With Sclerotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, Director of Vascular Surgery in ChengduUTCM, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChengduUTCMvs4
Record Dates: First submitted 2022-11-22; First posted 2022-12-16 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Vascular Diseases, Peripheral; Venous Insufficiency of Leg; Varicose Veins of Lower Limb
Keywords: Radiofrequency ablation combined with sclerotherapy; varicose veins; Sulodexide
MeSH Terms: conditions — Peripheral Vascular Diseases; Varicose Veins | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Intervention Model Description: A total of 120 patients with varicose veins who received radiofrequency ablation combined with sclerotherapy were randomly divided into two groups。 Each group included 60 people, one group added sulodexide based on the conventional treatment process, and the other group was a control group. The recovery of adverse reactions after surgery in both groups was observed.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taking sulodexide (Experimental): Sixty patients with varicose veins who received radiofrequency ablation combined with sclerotherapy were given Sulodexide softgels 250LSU twice a day for two months after surgery。
  Interventions: Drug: Sulodexide
- Not taking drug (No Intervention): Sixty patients with varicose veins of the lower extremities who received radiofrequency ablation combined with sclerotherapy were selected and did not take sulodexide after surgery.

INTERVENTIONS:
Drug: Sulodexide — The recovery of pigmentation, fibrosis, pain and other indicators in the group taking sulodexide after surgery, one month after surgery and three months after surgery was observed
  Arms: Taking sulodexide

SUMMARY:
The purpose of this study is to evaluate whether adding sulodexide to the patients with varicose veins who received radiofrequency ablation combined with sclerotherapy can reduce or improve the impact of adverse events。

DETAILED DESCRIPTION:
Chronic venous insufficiency（CVI）of the lower extremities is a commonly clinically syndrome。 It can manifest as telangiectasias (or spider veins), reticular veins, varicose veins（VVS）, edema, pigmentation and/or eczema, liposomal sclerosis, white atrophy, and venous ulcers。 Patients often seek treatment for varicose veins because of cosmetic problems, pain, swelling, itching, ulcers, and other symptoms。 With the development of society, more and more patients require to choose local anesthesia, minimally invasive, and rapid recovery surgery. Radiofrequency ablation(RFA) combined with sclerotherapy is a treatment with a broad clinically applicable spectrum for varicose veins, ranging from the Great saphenous vein （GSV）trunk to telangiectases (or spider veins).US guidelines for treating varicose veins and chronic venous disease of the lower extremities recommend endovascular thermal ablation (including RFA) as safe and effective for treating saphenous venous insufficiency. Foam sclerotherapy is to close the diseased vein by mixing sclerosants with air in a particular proportion and injecting it into the venous blood vessels so that the vein generates artificial thrombus and fibrosis. Because of its simple, economical, and minimally invasive characteristics, it is widely used in clinical practice.

Pigmentation, fibrous induration, and pain are the most common complications after RFA combined with sclerotherapy. Hyperpigmentation is a brownish discoloration of the skin due to extravasation of red blood cells and hemosiderin deposition。 Fibrous induration and pain are mainly caused by thrombosis, inflammation, and vascular fibrosis。 Sulodexide is an orally vasoactive drug consisting of 80% heparin sulfate + 20% corn sulfate， with antithrombotic, fibrinolytic, anti-inflammatory, endothelial protective, and vascular regulating properties. This agent is used in venous ulcers, prevents recurrent venous thromboembolism, and has a low incidence of bleeding complications.

Clinical observation in our department found that adding sulodexide can reduce or improve the impact of adverse events after RFA combined with sclerotherapy。

The purpose of this study is to evaluate whether adding sulodexide to the patients with varicose veins who received RFA combined with sclerotherapy accelerates the dissipation of pigmentation and fibrosis。

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <80 years, and able to understand the requirements of the study and provide informed consent and accept the exams and follow-up.
* C2 - C5 varicose veins / CVI Symptomatic primary GSV, SSV, or AASV incompetence, with reflux >0.5 seconds on color duplex, eligible for patients undergoing radiofrequency ablation plus sclerotherapy
* BMI<35
* The skin color is within the normal range, and no obvious skin color unevenness or skin diseases affect the observed indicators.

Exclusion Criteria:

* Acute superficial or deep vein thrombosis
* History of asthma and stroke
* There are skin diseases, scars, infections, and other conditions in the surgical area that affect the observation indicators
* Pregnancy
* Serious damage to liver and kidney function
* Severe obesity (BMI>35) and severe edema of the lower extremities
* Others are not eligible for intravenous radiofrequency ablation combined with sclerotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in pigmentation area and color depth over the three months after surgery. | three months
  Computer software（ImageJ and Brown pixel distribution histogram joint color deconvolution） is used to calculate and record the area of pigmentation and color depth and compare them at different times.
Changes in the incidence and hardness (Shore hardness) of fibrous induration in the three months after surgery. | three months
  The hardness of the fiber induration is calculated and recorded using a Shore hardness tester and compared at different times.The hardness should decrease as the hard knot softens。
Changes in the area of congestion in the three months after surgery. | three months
  Computer software（ImageJ） calculates and records the area of congestion and compares it at different times.

SECONDARY OUTCOMES:
Changes in pain scores on a visual analogue scale over the three months postoperatively postoperative | three months
  Pain scores are recorded on a Visual Analogue Scale and compared at different times.The scale ranges from 1 to 10, and the higher the score, the more painful it is
Incidence of bleeding complications | three months
  Regularly review and follow up with patients for the incidence of bleeding complications.（Such as hematemesis, vomiting blood, melena, etc）

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China